CLINICAL TRIAL: NCT04847128
Title: The Effect of Exercise on Anxiety and Cognition in Students at University: A Randomized Controlled Trial
Brief Title: The Effect of Exercise on Anxiety and Cognition in Students at University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XJTU1AF2020LSK-276
Record Dates: First submitted 2021-04-06; First posted 2021-04-19 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Exercise; Anxiety; Depression; Cognition
MeSH Terms: conditions — Motor Activity; Anxiety Disorders; Depression | interventions — Post-Exercise Recovery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors and statisticians were blinded to group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Participants receive exercise intervention 3 times weekly for 8 weeks.
  Interventions: Behavioral: Chronic aerobic exercise
- Arm II (No Intervention): Participants keep sedentary life without exercise for 8 weeks.

INTERVENTIONS:
Behavioral: Chronic aerobic exercise — Participants in the experimental group will exercise more than 30 minutes each time and 3 times weekly for 8 weeks. The chronic aerobic exercise in the present trial is running. The heart rate is required to 60% -85% of the maximum heart rate during exercise. Maximum heart rate = 220 - age.
  Other Names: Workout
  Arms: Arm I

SUMMARY:
RATIONALE: Exercise may improve the mood and cognition in young people.

PURPOSE: It has been well-known that physical exercise can generally benefit the mental health. However, most evidences that physical exercise improves psychiatric symptoms come from retrospective or cross-sectional studies. Moreover, the studies on the effect of physical exercise in the young adults' mental health were limited. This randomized-controlled trial aims to determinate the effects of a chronic and aerobic exercise on the mood and cognition of young people.

DETAILED DESCRIPTION:
OBJECTIVES: The anxiety and depression symptoms in young people are worth paying attention to, in China and worldwide. Meanwhile, cognitive function is very important for young people's learning and work. This project aims to evaluate the effectiveness of the moderate aerobic exercise to alleviate anxiety and depression in young people.

DESIGN & METHODS: Undergraduate and graduate students aged 18-35 years will be randomly and evenly assigned to exercise and control groups. Subjects assigned to exercise group will receive an running exercise intervention more than 30 minutes and 3 times per week for 8 weeks. The control group will be advised not to engage in physical activities. Outcome measures include the score of the Self-rating Anxiety Scale (SAS), Self-rating Depression Scale (SDS), the response time of Schulte Grid test, and the response time of Stroop Colour-Word Test at baseline and post-intervention in two groups. In addition, these assessments will be followed up at week 20 (3 months after the end of intervention).

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate and graduate students aged 18 to 35 years.

Exclusion Criteria:

* Heart disease, hypertension, cardiovascular and respiratory system diseases such as asthma and are unable to tolerate the frequency and strength of exercise requirements.
* Any neurological or psychiatric disorders.
* Physical disabilities.
* Severe dysmenorrhea when they couldn't exercise more than 5 days before or after menstruation.
* Color blindness.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2022-01-09 (Actual)

PRIMARY OUTCOMES:
Changes in the Self-rating Anxiety Scale (SAS) after intervention and at follow-up | Change from baseline to post-intervention at week 8 and follow up (3 months after intervention)
  The SAS is organized in 20 items, each with a score from 1 to 4, and a total score from 20 to 80. It will report the anxious mood, physical symptoms, psychomotor behavior and psychological symptoms of participants. Higher scores on the SAS indicate a higher level of anxiety symptoms.

SECONDARY OUTCOMES:
Changes in the Self-rating Depression Scale (SDS) after intervention and at follow-up | Change from baseline to post-intervention at week 8 and follow up (3 months after intervention)
  The SDS scale is organized in 20 items, each with a score from 1 to 4, and a total score from 20 to 80. It will report the depressive mood, physical symptoms, psychomotor behavior and psychological symptoms of participants. Higher scores on the SDS indicate a higher level of depressive symptoms.
Changes in the response times of Schulte Grid after intervention and at follow-up | Change from baseline to post-intervention at week 8 and follow up (3 months after intervention)
  In Schulte Grid test, the participants will be asked to point out randomly arranged 36 numbers within a 6 × 6 matrix in ascending order. Shorter time to finish the Schulte Grid test indicates a higher level of attention and cognition.
Changes in the response time of the Stroop Colour-Word Test after intervention and at follow-up | Change from baseline to post-intervention at week 8 and follow up (3 months after intervention)
  In Stroop Colour-Word test, the participants will be required to naming the colour of words printed in conflicting ink colours while refraining from reading the words (e.g., the word 'green' printed in blue ink). It measures cognitive control and inhibition of concurrent automatic process of word reading, both of which relate to executive functions. Participants will be instructed to name the colour while refraining from reading the words. The response times will be recorded to evaluate the level of attention and cognition.

OTHER OUTCOMES:
Alterations of sera proteome | week 8
  Using a proteomic analysis to compare the levels of proteins in the serum of participants between two groups after an 8-week exercise intervention.
Alterations of gut microbiota | week 8
  Using a shotgun metagenomic analysis to identify the alterations of gut microbiota in participants between two groups of after an 8-week exercise intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, MD., PhD., Principal Investigator — First Afflicated Hospital Xian Jiaotong University
Locations (1):
- First Afflicated Hospital Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
After 12/01/2023, by email requirement
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12/01/2023
Access Criteria: For scientific research only, not for commercial use

REFERENCES:
- [Background] Christiansen L, Beck MM, Bilenberg N, Wienecke J, Astrup A, Lundbye-Jensen J. Effects of Exercise on Cognitive Performance in Children and Adolescents with ADHD: Potential Mechanisms and Evidence-based Recommendations. J Clin Med. 2019 Jun 12;8(6):841. doi: 10.3390/jcm8060841. PMID 31212854
- [Background] Pedersen BK, Febbraio MA. Muscles, exercise and obesity: skeletal muscle as a secretory organ. Nat Rev Endocrinol. 2012 Apr 3;8(8):457-65. doi: 10.1038/nrendo.2012.49. PMID 22473333
- [Background] Lourenco MV, Frozza RL, de Freitas GB, Zhang H, Kincheski GC, Ribeiro FC, Goncalves RA, Clarke JR, Beckman D, Staniszewski A, Berman H, Guerra LA, Forny-Germano L, Meier S, Wilcock DM, de Souza JM, Alves-Leon S, Prado VF, Prado MAM, Abisambra JF, Tovar-Moll F, Mattos P, Arancio O, Ferreira ST, De Felice FG. Exercise-linked FNDC5/irisin rescues synaptic plasticity and memory defects in Alzheimer's models. Nat Med. 2019 Jan;25(1):165-175. doi: 10.1038/s41591-018-0275-4. Epub 2019 Jan 7. PMID 30617325
- [Background] Moon HY, Becke A, Berron D, Becker B, Sah N, Benoni G, Janke E, Lubejko ST, Greig NH, Mattison JA, Duzel E, van Praag H. Running-Induced Systemic Cathepsin B Secretion Is Associated with Memory Function. Cell Metab. 2016 Aug 9;24(2):332-40. doi: 10.1016/j.cmet.2016.05.025. Epub 2016 Jun 23. PMID 27345423
- [Background] Horowitz AM, Fan X, Bieri G, Smith LK, Sanchez-Diaz CI, Schroer AB, Gontier G, Casaletto KB, Kramer JH, Williams KE, Villeda SA. Blood factors transfer beneficial effects of exercise on neurogenesis and cognition to the aged brain. Science. 2020 Jul 10;369(6500):167-173. doi: 10.1126/science.aaw2622. PMID 32646997
- [Background] Rosenberg MD, Finn ES, Scheinost D, Papademetris X, Shen X, Constable RT, Chun MM. A neuromarker of sustained attention from whole-brain functional connectivity. Nat Neurosci. 2016 Jan;19(1):165-71. doi: 10.1038/nn.4179. Epub 2015 Nov 23. PMID 26595653
- [Background] Ng QX, Ho CYX, Chan HW, Yong BZJ, Yeo WS. Managing childhood and adolescent attention-deficit/hyperactivity disorder (ADHD) with exercise: A systematic review. Complement Ther Med. 2017 Oct;34:123-128. doi: 10.1016/j.ctim.2017.08.018. Epub 2017 Aug 31. PMID 28917364
- [Background] de Greeff JW, Bosker RJ, Oosterlaan J, Visscher C, Hartman E. Effects of physical activity on executive functions, attention and academic performance in preadolescent children: a meta-analysis. J Sci Med Sport. 2018 May;21(5):501-507. doi: 10.1016/j.jsams.2017.09.595. Epub 2017 Oct 10. PMID 29054748